CLINICAL TRIAL: NCT04052815
Title: Culturally Adapted Community-based Translational Diabetes Prevention Program for Obese and Pre-diabetic Hispanic/Latino Females
Brief Title: Community Based DPP Program for Hispanic/Latino Females
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Nallely Mora, Research Assistant Professor, Loyola University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 212259
Record Dates: First submitted 2019-08-06; First posted 2019-08-12 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Pre Diabetes; Obesity
Keywords: pre-diabetes; female; Diabetes type 2; Hispanic/Latino; community based programs; diabetes prevention program
MeSH Terms: conditions — Glucose Intolerance; Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diabetes prevention program culturally tailored (Experimental): Adult females with Hispanic background
  Interventions: Behavioral: Diabetes prevention program culturally tailored

INTERVENTIONS:
Behavioral: Diabetes prevention program culturally tailored — Diabetes prevention Program (DPP) as specified by the CDC, physical activity prior to DPP sessions, motivational interviewing individual and in group. Culturally tailored nutrition tips and recipes.

SUMMARY:
Is well known that obesity is increasing in the United States (US) and particularly among Hispanic/ especially in in socially disadvantaged groups. Studies have shown that the prevalence of metabolic syndrome is about 1.5 times higher among Mexican American females living in the US compared to non-Hispanic females. Culturally among Hispanic/Latino females some activities like grocery shopping and meal cooking in households that most likely impact other family members.

Culturally grounded interventions can be made readily tailored and translated into real-world settings by utilizing collaborative, community based participatory approaches. The overall objective of this study is to offer a diabetes prevention program to the community, targeting adult females with Hispanic/Latino background population that could benefit from a sustainable change behavior program to reduce the risk of developing Type 2 Diabetes, metabolic syndrome and cardiovascular disease. Sessions will be conducted in Spanish or English according to participants' preferences. The program format is to meet for one year. Cadence will be once a week for the next 16 weeks (Core curriculum), then once a month (maintenance curriculum). In addition to the DPP curriculum a structured physical activity component will be added, with the objective of facilitating achievement of program goals. Other culturally tailored activities will be included like: grocery shopping, recipes community walking maps and other available community resources.

In addition the investigators will utilize a qualitative approach to gather information about project's feasibility and acceptability. To do so, investigators plan to conduct 60 minutes focus groups and semi structured interviews at the end of the 16 week core-program and at the end of the program (program participants and staff members).

DETAILED DESCRIPTION:
Is well known that obesity is increasing in the United States (US) and particularly among Hispanic/Latinos and African American women especially in in socially disadvantaged groups. Similarly, diabetes mellitus is a health care burden in the US, with associated costs estimated in $174 billion in 2007, and projections for 2030 estimate that about 30 million Americans will have diabetes. Studies have shown that the prevalence of metabolic syndrome is about 1.5 times higher among Mexican American females living in the US compared to non-Hispanic females.

Latinos is one of the largest ethnic groups in the Chicago metropolitan region, in Cook county they comprise about 25% of the population (around 1,295,000 people), and of those 75% are of Mexican origin followed by Puerto Rican (13%).

In addition 17% of the population in Chicagoland area does not count with health insurance, the Latino community having the higher percent of uninsured population ranging from 18-32%. This puts in disadvantage the Hispanic/Latino population with high risk factors to develop chronic diseases that have proven to be more prevalent amongst them, like T2D and metabolic syndrome. Culturally among Hispanic/Latino females some activities like grocery shopping and meal cooking in households that most likely impact other family members.

Culturally grounded interventions can be made readily tailored and translated into real-world settings by utilizing collaborative, community based participatory approaches. From a public health perspective, these approaches may offer the greater likelihood for closing the obesity related health disparities gap that currently exist among community members in the US population.

The Diabetes Prevention Program (DPP), a randomized controlled trial of a lifestyle change program implemented from 1996 through 2002 with up to 5 years of follow up, demonstrated that individuals with prediabetes who achieved between 5-7% weight reduction and participated in regularly physical activity reduced their T2D risk between 58-71%, twice that achieved through medication. Specifically the DPP program has two main goals: weight loss through healthy eating, aiming for 5-7%; and regular physical activity (PA) to improve overall health, aiming for 150 minutes of brisk PA per week. The program is delivered over a year by DPP trained lifestyle coaches.

Community-based lifestyle interventions (CBLI) have been proposed as an effective mechanisms to improve the health of local communities through health education and the adoption of healthier behaviors. This community approach rests on the premise that the intervention respects community strengths, is dictated by cultural practices, and depends on meaningful community participation.

The overall objective of this study is to offer a diabetes prevention program in one of the nearby communities to Loyola University Health System, targeting a minority population that could highly benefit from a sustainable change behavior program to reduce the risk of developing T2D, metabolic syndrome and cardiovascular disease among identified high risk individuals. Towards these end, the investigators proposed a community based translational diabetes prevention program, and qualitative research methods to evaluate its acceptability, feasibility and effectiveness. This study will used a mixed research methods approach. For each aim the investigators proposed the following methods:

Aim1: Implementation of a Pilot Diabetes prevention program targeting Hispanic/Latino females with obesity or pre-diabetes in nearby communities.

* The investigators will hold community health fairs to increase awareness among community stakeholders and community members about the existence of prevention programs that could benefit their health at long term. The aim is to drive from this events potential participants for the pilot program.
* The one year long diabetes Prevention program developed by the CDC will be delivered as prescribed in preferred language, which investigators assumed will be Spanish. In addition to the DPP curriculum a structured physical activity component will be added, with the objective of facilitating achievement of program goals. Nutrition education will be delivered focused on traditional Latino foods. In addition to the CDC original DPP the investigators will give a pedometer to each participant, include organized weekly physical activity sessions, community walking maps, and resources in which at low cost participants will be able to reach the program 150 min/week PA goal. Additional reinforcement activities out of class will be offered such as grocery shopping with family members to prepare a healthy family meal, food demonstrations, recipes related to themes will facilitate curriculum integration into day-to-day lifestyle changes.

Aim2: Assess the acceptability in this specific community for a community based translational diabetes prevention program.

•After 16 weeks of program start, the investigators will carry out focus groups with participants, and semi-structured interviews with lifestyle coaches and key community stakeholders, with the intention to improve program planning and delivery for the next cycle-2020.

Aim 3: Gather preliminary data about feasibility and potential effectiveness of a community based translational diabetes prevention program for Hispanic/Latino females in a community setting.

•At program conclusion the investigators will carry out a second round of focus groups with participants, and semi-structured interviews with lifestyle coaches. The objective is to learn about barriers and success stories from lifestyle coaches, research team and community members that faced during the different phases of the program. Feedback from program facilitators and participants will help to seek opportunities to improve community based DPP program delivery.

ELIGIBILITY:
Inclusion Criteria:

* Hispanic/Latino background, female, ≥18 years old, with Body mass index (BMI) ≥25 or Glycated hemoglobin (Hb1AC) and/or glucose on parameter to be considered pre-diabetic.

Exclusion Criteria:

* to have a diagnosis of diabetes, taking medication for diabetes, conditions that impedes mobilization, mental impairment, or conditions that impede to be under diet restrictions.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Weight at 12 month | 12 months
  weight in lb
Change from Baseline waist circumference at 12 months | 12 months
  waist circumference in centimeters
Change from Baseline Glycated hemoglobin at 12 months | 12 months
  Glycated hemoglobin (HbA1C)

SECONDARY OUTCOMES:
Change from Baseline low density lipoprotein (LDL) at 12 months | 12 months
  low density lipoprotein
Change from baseline High-density lipoprotein (HDL) at 12 months | 12 months
  High-density lipoprotein
Dietary assessment for fruits and vegetables | baseline, 16 weeks, 12 months
  Dietary assessment for fruits and vegetables using a score in which the first-administration times-per-day score on the simple score yielded the following equations Fruit and vegetables times/day=0.34+ Fruit/vegetable simple-1.34. The score obtained could be interpreted as: <13 equals poor, 13-15 =fair, 16-17= good and =>18 excellent. The screener is in relation to the past month consumption of vegetables and fruits and how often do they consume per week a product
Dietary assessment of fat consumption | baseline, 16 weeks, 12 months
  Dietary assessment of fat consumption The screener is in relation to the past month consumption of fat and how often do they consume per week a product. Scale construct is the first-administration times-per-day score on the simple score yielded the following equations Fat Times/day= 0.16+fat simple-0.48. The score obtained could be interpreted as: =< 18-excellent, 19-24-good, 25-33-fair, >33-poor

OTHER OUTCOMES:
7-day physical activity recall | baseline, 16 weeks, 12 months
  Recall instrument that measures the type of physical activity performed during the past 7 days
Perceived self-efficacy | baseline, 16 weeks, 12 months
  Perceived self-efficacy by Schwarzer. The total score is calculated by finding the sum of the all items. For the General Self Efficacy, the total score ranges between 10 and 40, with a higher score indicating more self-efficacy
Rosenberg self-esteem | baseline and 12 months
  self report measure that pertain self-worth and self acceptance. Rated on a 4-point Likert-type scale, ranging from 1 (totally disagree) to 4 (totally agree). Items 1, 3, 4, 7, and 10 are positively worded, and items 2, 5, 6, 8, and 9 negatively. Sum scores for all ten items. Keep scores on a continuous scale. Higher scores indicate higher self-esteem.

CONTACTS AND LOCATIONS:
Overall Officials: Nallely Mora, MD, MPH, Principal Investigator — Loyola University Chicago
Locations (1):
- Quinn Center, Maywood, Illinois, United States

REFERENCES:
- [Background] Wyatt SB, Winters KP, Dubbert PM. Overweight and obesity: prevalence, consequences, and causes of a growing public health problem. Am J Med Sci. 2006 Apr;331(4):166-74. doi: 10.1097/00000441-200604000-00002. PMID 16617231
- [Background] Wild S, Roglic G, Green A, Sicree R, King H. Global prevalence of diabetes: estimates for the year 2000 and projections for 2030. Diabetes Care. 2004 May;27(5):1047-53. doi: 10.2337/diacare.27.5.1047. PMID 15111519
- [Background] Ervin RB. Prevalence of metabolic syndrome among adults 20 years of age and over, by sex, age, race and ethnicity, and body mass index: United States, 2003-2006. Natl Health Stat Report. 2009 May 5;(13):1-7. PMID 19634296
- [Background] Acosta-Cordova, The Latino Neighborhood report: issues and prospects for Chicago. Institute for research on race and public policy, Great city Institute, University of Illinois at Chicago. , 2017.
- [Background] Arbona C, Olvera N, Rodriguez N, Hagan J, Linares A, Wiesner M. Acculturative Stress Among Documented and Undocumented Latino Immigrants in the United States. Hisp J Behav Sci. 2010 Aug;32(3):362-384. doi: 10.1177/0739986310373210. PMID 25484488
- [Background] Shobe MA, Coffman MJ, Dmochowski J. Achieving the American dream: facilitators and barriers to health and mental health for Latino immigrants. J Evid Based Soc Work. 2009 Jan;6(1):92-110. doi: 10.1080/15433710802633601. PMID 19199139
- [Background] Katy M. Pinto, V.O., Beyond Cultural Explanations: Understanding the Gendered Division of Household Labor in Mexican American Families. Journal of Family Issues, 2018. 39(16).
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Centers for Disease, C.a.P., Diabetes prevention Recognition program: standards and operating procedures, Atlanta (GA). US Department of Health and Human Services, 2011.
- [Background] Satterfield DW, Volansky M, Caspersen CJ, Engelgau MM, Bowman BA, Gregg EW, Geiss LS, Hosey GM, May J, Vinicor F. Community-based lifestyle interventions to prevent type 2 diabetes. Diabetes Care. 2003 Sep;26(9):2643-52. doi: 10.2337/diacare.26.9.2643. PMID 12941733
- [Background] Viswanathan M, Ammerman A, Eng E, Garlehner G, Lohr KN, Griffith D, Rhodes S, Samuel-Hodge C, Maty S, Lux L, Webb L, Sutton SF, Swinson T, Jackman A, Whitener L. Community-based participatory research: assessing the evidence. Evid Rep Technol Assess (Summ). 2004 Aug;(99):1-8. No abstract available. PMID 15460504
- [Background] Wallerstein N, Duran B. Community-based participatory research contributions to intervention research: the intersection of science and practice to improve health equity. Am J Public Health. 2010 Apr 1;100 Suppl 1(Suppl 1):S40-6. doi: 10.2105/AJPH.2009.184036. Epub 2010 Feb 10. PMID 20147663
- [Background] Wakimoto P, Block G, Mandel S, Medina N. Development and reliability of brief dietary assessment tools for Hispanics. Prev Chronic Dis. 2006 Jul;3(3):A95. Epub 2006 Jun 15. PMID 16776896